CLINICAL TRIAL: NCT03300297
Title: Thrust Joint Manipulation to the Cervical Spine in Participants With a Primary Complaint of Temporomandibular Disorder (TMD): A Randomized Clinical Trial
Brief Title: Cervical Spine Thrust Joint Manipulation for Temporomandibular Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley University (Other)
Collaborators: Nova Southeastern University (Other); University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Breanna Reynolds, Assistant Professor, Bradley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BU 59-16
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular joint; Physical Therapy; Cervical spine thrust joint manipulation; therapy, exercise; Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention groups. Both will receive intervention and one group will receive cervical spine thrust joint manipulation while the other receives sham manipulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation. Blind assessors will be utilized to measure objective change in range of motion and pain pressure threshold.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Spine Thrust Joint Manipulation (Active Comparator): Thrust Manipulation delivered to C0/1 and C2/3 on both the right and left side
  Interventions: Other: Cervical Spine Thrust Joint Manipulation; Other: Home Program; Other: Suboccipital Release
- Cervical Spine Sham Manipulation (Sham Comparator): Sham Manipulation delivered to C0/1 and C2/3 on both the right and left side
  Interventions: Other: Cervical Spine Sham Manipulation; Other: Home Program; Other: Suboccipital Release

INTERVENTIONS:
Other: Cervical Spine Thrust Joint Manipulation — High velocity, short amplitude thrust to the cervical spine
  Other Names: Grade V manipulation
  Arms: Cervical Spine Thrust Joint Manipulation
Other: Cervical Spine Sham Manipulation — Manipulative hold position shy of end range without a thrust
  Arms: Cervical Spine Sham Manipulation
Other: Home Program — therapeutic exercise program and education
Other: Suboccipital Release — suboccipital soft tissue mobilization
  Other Names: soft tissue mobilization

SUMMARY:
Background: Temporomandibular disorder (TMD) is a common and costly problem that often leads to chronic pain or dysfunction. There is moderate evidence to support physical therapy (PT) interventions for individuals with TMD, yet they continue to be an underserved population. A known relationship between TMD and the cervical spine exists with some evidence to support the use of cervical interventions for TMD. Cervical spine thrust joint manipulation (TJM) is an effective PT intervention that has been explored in a limited fashion for this population.

The purpose of this trial is to determine the immediate and short term (1 and 4 week) effects of cervical TJM delivered by a physical therapist on pain, dysfunction, and perception of change in persons with a primary complaint of TMD. The hypothesis is that all participants will improve, and those in the cervical TJM group may have a greater degree of improvement.

Design: Participants will be randomized to one of two groups and all will receive physical therapy. Forty-two willing participants, age 18-65 with TMD will complete the informed consent process and screening for eligibility before being admitted. Participants will receive a combined treatment of 1) behavioral education, a home exercise program, soft tissue mobilization, and cervical spine TJM or 2) behavioral education, a home exercise program, soft tissue mobilization, and sham manipulation. Participants will receive 4 treatments over a period of 4 weeks.

Significance: The results of this clinical trial will provide evidence relative to the impact of cervical spine TJM in the treatment of persons with TMD. Determining the effectiveness of cervical spine TJM included with a combined treatment approach has clinical implication for physical therapists and the patients they serve.

DETAILED DESCRIPTION:
Methods: Research design following CONSORT guidelines. A blinded assessor will measure ROM and PPT. Treating therapists will know group allocation and will receive training to standardize assessments and treatments. Self-report and objective measurements will be taken at baseline, immediately after treatment one, and at one and four week follow-ups.

Data Analysis (primary): Sample size estimations were completed using G-Power, a free online downloadable program. An F-test family with ANOVA: Repeated measures, within-between interaction protocol was selected. While it is optimal to power sample size estimations around a functional outcome measure, the limited use of functional measures in this population created an obstacle. The sample size estimation for this project was powered around maximal mouth opening (MMO) as this most closely relates to function in the TMD population. In order to account for 15% attrition, and maintain equal participants in each arm of this study, the desired sample size is 42 participants.

A 2 x 4 mixed model analysis of variance (ANOVA) will be used with treatment group as the between-subjects factor and time as the within-subjects factor. Separate ANOVAs will be performed for dependent variables and the hypothesis of interest will be group by time interaction for each ANOVA.

To determine if missing data points associated with dropouts were missing at random or missing for systematic reasons, we will perform Little's Missing Completely at Random (MCAR) Test. Intention to treat analysis will be performed by using expectation maximization whereby missing data are computed using regression equations. Planned pair-wise comparisons will examine the difference between baseline and follow-up periods using the Bonferroni equality at an alpha level of 0.05.

Success will be dichotomized using the GROC scale. A cut-off score of +5 or higher on the GROC will be used as a measure of success. Correlations between outcome measures (change scores) and success will be analyzed using an independent t-test to determine if differences between groups exist. Number needed to treat (NNT) will be calculated. Correlations among dependent variables will be analyzed with Pearson/Spearman correlations. Examples include the following: correlation between NDI and jaw functional measures, correlation among PPT at various areas tested, and correlation between change in ROM and change in functional scores. Data analysis will include 95% confidence intervals, and tables, charts, or other figures will be utilized to display findings to enhance reader understanding. Effect size of primary outcome measures including jaw ROM, JFLS, and TMD Disability Index will be calculated and reported. If there is no significant difference between groups noted, a post-hoc power analysis will be performed to determine the risk of Type II error.

Data Safety Plan/Subject Confidentiality: The PI will be responsible for educating all clinicians, research assistants, and front office staff with RVPT, Bradley University, and UNLV in confidentiality measures and data safety plans. This information will be part of the live training and included in the Manuals of Standard Operating Procedures. The PI will also periodically check in with each participating clinician, blinded assessor, and clinic office staff member to review procedures and monitor recruitment and retention. This check will occur once per month over the phone.

Standard Operating Procedures: Manual developed and used in training.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 y/o
* primary complaint of TMD pain
* positive TMD screen
* proficiency in English language
* availability to attend 4 sessions
* minimum level of disability (NPRS 2 or greater)
* minimum level of disability (pain free mouth opening 50 mm or less).

Exclusion Criteria:

* traumatic onset of symptoms
* whiplash in the last 6 weeks
* prior neck surgery
* medical red flags suggestive on on-musculoskeletal origin of pain, systemic disease, or neurological disease
* contraindications to thrust joint manipulation (TJM),
* previous TJM in the last 3 months
* Worker's compensation
* pending litigation regarding pain or injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Maximal Mouth Opening Range of Motion (mm) | baseline, immediate, 1 week, 4 week
  Jaw ROM, mouth opening
Change in Pain with Numeric Pain Rating Scale | baseline, immediate, 1 week, 4 week
  NPRS, self-reported intensity of pain on 0-10 pain rating scale
Change in Function with Jaw Functional Limitation Scale | baseline, 1 week, 4 week, 3 month, 6 month
  JFLS, self report jaw functions rated 0-10 based on difficulty
Change in Fear with Tampa Scale of Kinesiophobia-TMD version | baseline, 1 week, 4 week, 3 month, 6 month
  self report scale to assess level of fear rating 12 items on a 1-4 scale
Global Rating of Change | immediate, 1 week, 4 week
  perception of overall change in a self report scale from -7 to +7

SECONDARY OUTCOMES:
Change in Function with Neck Disability Index | baseline, 1 week, 4 week, 3 month, 6 month
  10 item self report assessment of neck disability
Change in Function with TMD Disability Index | baseline, 1 week, 4 week, 3 month, 6 month
  10 item self report assessment of jaw dysfunction
Patient Acceptable Symptom State | 4 week, 3 month, 6 month
  Self report acceptable nature of current state
Change in Cervical Spine range of motion | baseline, immediate, 1 week, 4 week
  bubble inclinometer measurement of neck motion
Change in Pain pressure threshold | baseline, immediate, 1 week, 4 week
  digital algometer assessment of threshold
PHQ-2 Depression Screen | baseline
  2 question screen

CONTACTS AND LOCATIONS:
Overall Officials: Breanna C Reynolds, DPT, Principal Investigator — Bradley University
Locations (2):
- United States (2):
  - Rock Valley Physical Therapy, Peoria, Illinois
  - Rock Valley Physical Therapy, Washington, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Harrison AL, Thorp JN, Ritzline PD. A proposed diagnostic classification of patients with temporomandibular disorders: implications for physical therapists. J Orthop Sports Phys Ther. 2014 Mar;44(3):182-97. doi: 10.2519/jospt.2014.4847. PMID 24579796
- [Background] Kraus SL. Characteristics of 511 patients with temporomandibular disorders referred for physical therapy. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Oct;118(4):432-9. doi: 10.1016/j.oooo.2014.06.005. Epub 2014 Jul 2. PMID 25240990
- [Background] Martins WR, Blasczyk JC, Aparecida Furlan de Oliveira M, Lagoa Goncalves KF, Bonini-Rocha AC, Dugailly PM, de Oliveira RJ. Efficacy of musculoskeletal manual approach in the treatment of temporomandibular joint disorder: A systematic review with meta-analysis. Man Ther. 2016 Feb;21:10-7. doi: 10.1016/j.math.2015.06.009. Epub 2015 Jun 25. PMID 26144684
- [Background] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Background] McNeely ML, Armijo Olivo S, Magee DJ. A systematic review of the effectiveness of physical therapy interventions for temporomandibular disorders. Phys Ther. 2006 May;86(5):710-25. PMID 16649894
- [Background] Paco M, Peleteiro B, Duarte J, Pinho T. The Effectiveness of Physiotherapy in the Management of Temporomandibular Disorders: A Systematic Review and Meta-analysis. J Oral Facial Pain Headache. 2016 Summer;30(3):210-20. doi: 10.11607/ofph.1661. PMID 27472523
- [Background] Silveira A, Gadotti IC, Armijo-Olivo S, Biasotto-Gonzalez DA, Magee D. Jaw dysfunction is associated with neck disability and muscle tenderness in subjects with and without chronic temporomandibular disorders. Biomed Res Int. 2015;2015:512792. doi: 10.1155/2015/512792. Epub 2015 Mar 26. PMID 25883963
- [Background] Olivo SA, Fuentes J, Major PW, Warren S, Thie NM, Magee DJ. The association between neck disability and jaw disability. J Oral Rehabil. 2010 Sep;37(9):670-9. doi: 10.1111/j.1365-2842.2010.02098.x. Epub 2010 May 27. PMID 20524969
- [Background] La Touche R, Fernandez-de-las-Penas C, Fernandez-Carnero J, Escalante K, Angulo-Diaz-Parreno S, Paris-Alemany A, Cleland JA. The effects of manual therapy and exercise directed at the cervical spine on pain and pressure pain sensitivity in patients with myofascial temporomandibular disorders. J Oral Rehabil. 2009 Sep;36(9):644-52. doi: 10.1111/j.1365-2842.2009.01980.x. Epub 2009 Jul 14. PMID 19627454
- [Background] La Touche R, Paris-Alemany A, Mannheimer JS, Angulo-Diaz-Parreno S, Bishop MD, Lopez-Valverde-Centeno A, von Piekartz H, Fernandez-Carnero J. Does mobilization of the upper cervical spine affect pain sensitivity and autonomic nervous system function in patients with cervico-craniofacial pain?: A randomized-controlled trial. Clin J Pain. 2013 Mar;29(3):205-15. doi: 10.1097/AJP.0b013e318250f3cd. PMID 22874091
- [Background] Gonzalez YM, Schiffman E, Gordon SM, Seago B, Truelove EL, Slade G, Ohrbach R. Development of a brief and effective temporomandibular disorder pain screening questionnaire: reliability and validity. J Am Dent Assoc. 2011 Oct;142(10):1183-91. doi: 10.14219/jada.archive.2011.0088. PMID 21965492
- [Background] Kraus S. Temporomandibular disorders, head and orofacial pain: cervical spine considerations. Dent Clin North Am. 2007 Jan;51(1):161-93, vii. doi: 10.1016/j.cden.2006.10.001. PMID 17185065
- [Background] Medlicott MS, Harris SR. A systematic review of the effectiveness of exercise, manual therapy, electrotherapy, relaxation training, and biofeedback in the management of temporomandibular disorder. Phys Ther. 2006 Jul;86(7):955-73. PMID 16813476
- [Background] Calixtre LB, Moreira RF, Franchini GH, Alburquerque-Sendin F, Oliveira AB. Manual therapy for the management of pain and limited range of motion in subjects with signs and symptoms of temporomandibular disorder: a systematic review of randomised controlled trials. J Oral Rehabil. 2015 Nov;42(11):847-61. doi: 10.1111/joor.12321. Epub 2015 Jun 7. PMID 26059857
- [Background] Mansilla-Ferragut P, Fernandez-de-Las Penas C, Alburquerque-Sendin F, Cleland JA, Bosca-Gandia JJ. Immediate effects of atlanto-occipital joint manipulation on active mouth opening and pressure pain sensitivity in women with mechanical neck pain. J Manipulative Physiol Ther. 2009 Feb;32(2):101-6. doi: 10.1016/j.jmpt.2008.12.003. PMID 19243721
- [Background] Oliveira-Campelo NM, Rubens-Rebelatto J, Marti N-Vallejo FJ, Alburquerque-Sendi N F, Fernandez-de-Las-Penas C. The immediate effects of atlanto-occipital joint manipulation and suboccipital muscle inhibition technique on active mouth opening and pressure pain sensitivity over latent myofascial trigger points in the masticatory muscles. J Orthop Sports Phys Ther. 2010 May;40(5):310-7. doi: 10.2519/jospt.2010.3257. PMID 20436241
- [Background] Mulet M, Decker KL, Look JO, Lenton PA, Schiffman EL. A randomized clinical trial assessing the efficacy of adding 6 x 6 exercises to self-care for the treatment of masticatory myofascial pain. J Orofac Pain. 2007 Fall;21(4):318-28. PMID 18018993
- [Background] Armijo-Olivo S, Magee D. Cervical musculoskeletal impairments and temporomandibular disorders. J Oral Maxillofac Res. 2013 Jan 1;3(4):e4. doi: 10.5037/jomr.2012.3404. eCollection 2013. PMID 24422022
- [Background] La Touche R, Fernandez-de-Las-Penas C, Fernandez-Carnero J, Diaz-Parreno S, Paris-Alemany A, Arendt-Nielsen L. Bilateral mechanical-pain sensitivity over the trigeminal region in patients with chronic mechanical neck pain. J Pain. 2010 Mar;11(3):256-63. doi: 10.1016/j.jpain.2009.07.003. Epub 2009 Nov 27. PMID 19945351
- [Background] Calixtre LB, Gruninger BL, Haik MN, Alburquerque-Sendin F, Oliveira AB. Effects of cervical mobilization and exercise on pain, movement and function in subjects with temporomandibular disorders: a single group pre-post test. J Appl Oral Sci. 2016 May-Jun;24(3):188-97. doi: 10.1590/1678-775720150240. PMID 27383698
- [Background] Cuccia AM, Caradonna C, Annunziata V, Caradonna D. Osteopathic manual therapy versus conventional conservative therapy in the treatment of temporomandibular disorders: a randomized controlled trial. J Bodyw Mov Ther. 2010 Apr;14(2):179-84. doi: 10.1016/j.jbmt.2009.08.002. Epub 2009 Sep 20. PMID 20226365
- [Background] Visscher CM, Ohrbach R, van Wijk AJ, Wilkosz M, Naeije M. The Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD). Pain. 2010 Sep;150(3):492-500. doi: 10.1016/j.pain.2010.06.002. Epub 2010 Jul 3. PMID 20598804